CLINICAL TRIAL: NCT01794741
Title: Randomized Trial of the Safety of Dymista Nasal Spray and Fluticasone Propionate Nasal Spray in Children Ages >4 Years to <12 Years With Allergic Rhinitis
Brief Title: 3 Month Safety Study of Dymista Nasal Spray and Fluticasone Propionate in Children 4-11 Years of Age With Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP 4007
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Results first posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dymista nasal spray (Active Comparator): azelastine 137mcg per spray/fluticasone propionate 50mcg per spray one spray per nostril twice a day for three months
  Interventions: Drug: Dymista Nasal Spray
- fluticasone propionate nasal spray (Active Comparator): fluticasone propionate nasal spray 50mcg per spray per nostril twice a day
  Interventions: Drug: Fluticasone propionate nasal spray

INTERVENTIONS:
Drug: Dymista Nasal Spray
  Arms: Dymista nasal spray
Drug: Fluticasone propionate nasal spray
  Arms: fluticasone propionate nasal spray

SUMMARY:
This is a 3 month safety study of Dymista Nasal spray in children aged 4 to 11 years with allergic rhinitis

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 4 years to <12 years, inclusive at the screening visit
* A history of allergic rhinitis (AR)
* The parent/caregiver must provide written informed consent and the child must provide assent
* Willing and able to comply with the study requirements
* Require treatment with Dymista Nasal Spray, based on the Investigator's assessment (based on medical history, physical examination, etc.) of the subjects' clinical condition, at both the Screening and Randomization Visits
* General good health and free of any disease or concomitant treatment that could interfere with the interpretation of the study results as determined by the investigator or the sponsor's medical officer
* Subjects receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit (adjustments to regimen following a brief period of missed injections do not preclude participation)

Exclusion Criteria:

* On nasal examination, subjects with superficial nasal mucosal erosion, moderate nasal mucosal erosion, nasal mucosal ulceration, nasal septum perforation
* Nasal disease(s) likely to affect deposition of intranasal medication, such as acute or chronic sinusitis, rhinitis medicamentosa, clinically significant polyposis or clinically significant nasal structural abnormalities
* Nasal surgery or sinus surgery within the previous year
* The use of any investigational drug within 30 days prior to Visit 1. No investigational products are permitted for use during the conduct of this study
* Presence of any hypersensitivity to azelastine hydrochloride and/or fluticasone propionate or drugs similar to azelastine hydrochloride and/or fluticasone propionate
* Respiratory tract infections within two weeks prior to Visit 1.
* Subjects with significant pulmonary disease including asthma. Subjects with intermittent asthma who only require short-acting inhaled bronchodilators (not more often than twice per week) and who do not have nocturnal awakening as a result of asthma are eligible for enrollment
* Chronic obstructive sleep apnea syndrome (clinical diagnosis)
* Existence of any surgical or medical condition, which in the opinion of the investigator or sponsor's medical monitor, might significantly alter the absorption, distribution, metabolism, or excretion of study drug or that might significantly affect the subject's ability to complete this trial
* Clinically relevant abnormal physical findings or laboratory results which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures
* Family members of research center or private practice personnel who are directly involved in this study are excluded
* Members of the same family cannot enroll in the study at the same time.
* Subjects who have used medications or therapies that could interfere with safety evaluations (see Sections 4.0 and 5.0) and have not had the proper washouts from these medications or therapies
* Any behavioral condition which could affect subject's ability to accurately report symptoms to the caregiver such as developmental delay, attention deficit disorder, and autism
* Positive pregnancy test in female subjects ≥ 9 years of age
* Females who are pregnant or nursing practicing a medically acceptable method of contraception
* Subjects who fail to complete the symptom diary during the lead-in period, defined as missing data for >50% of entries

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 405 (Actual)
Dates: Start 2013-02; Primary Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ruiz, M.D., Study Director — Sponsor GmbH
Locations (41):
- United States (41):
  - Clinical Research Center of Alabama,LLC, Birmingham, Alabama
  - Little Rock Allergy and Asthma Clinical research Center, Little Rock, Alaska
  - West Coast Clinical Trials, Costa Mesa, California
  - Allergy & Asthma Care Center of So. Cal, Long Beach, California
  - Southern California Research, Mission Viejo, California
  - Allergy Associates Medical Group Inc, San Diego, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Cntr, San Jose, California
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, PC, Denver, Colorado
  - Asthma and Allergy Associates, PC, Pueblo, Colorado
  - Allergy and Asthma Care of Florida, Ocala, Florida
  - Atlanta Allergy and Asthma Clinic, Stockbridge, Georgia
  - Idaho Allergy, Eagle, Idaho
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Clinical Research Institute of Indiana, Indianapolis, Indiana
  - Family Allergy and Asthma Reserach, Louisville, Kentucky
  - Respiratory Medicine Research Institute of Michigan, Ypsilanti, Michigan
  - Clinical Reseacrh Institute, Minneapolis, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Clinical Research of the Ozarks,Inc, Warrensburg, Missouri
  - Midwest Allergy and Asthma Clinic, Omaha, Nebraska
  - The Asthma and Allergy Center, PC, Papillion, Nebraska
  - Atlantic Research Center, Ocean City, New Jersey
  - Asthma, Sinus & Allergy Centers, LLC, Warren Township, New Jersey
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Oklahoma Institute of Allergy and Asthma, Oklahoma City, Oklahoma
  - Baker Allergy Asthma & Dermatology Ctr LLC, Lake Oswego, Oregon
  - Allergy and Asthma Specialist PC, Blue Bell, Pennsylvania
  - National Allergy, Asthna & Urticaria Centers of Charleston Pa, Charleston, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associate, Upland, Pennsylvania
  - ADAC Research, PA, Greenville, South Carolina
  - AARA Research Center, Dallas, Texas
  - Texas Allergy Research Center, Dallas, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Paul H Ratner,MD, San Antonio, Texas
  - Live Oak Allergy and Asthma Clinic, San Antonio, Texas
  - Allergy Asthma Research Institute, Waco, Texas
  - Pediatric Allergy,Asthma and Immunology/Allergy& Asthma care of Waco, Waco, Texas

REFERENCES:
- [Derived] Berger W, Sher E, Gawchik S, Fineman S. Safety of a novel intranasal formulation of azelastine hydrochloride and fluticasone propionate in children: A randomized clinical trial. Allergy Asthma Proc. 2018 Mar 1;39(2):110-116. doi: 10.2500/aap.2018.39.4116. PMID 29490769

RESULTS

PARTICIPANT FLOW:
Groups:
- Dymista Nasal Spray: azelastine 137mcg per spray/fluticasone propionate 50mcg per spray one spray per nostril twice a day for three months
  Dymista Nasal Spray
- Fluticasone Propionate Nasal Spray: fluticasone propionate nasal spray 50mcg per spray per nostril twice a day
  Fluticasone propionate nasal spray
Period: Overall Study
Arm/Group | Dymista Nasal Spray | Fluticasone Propionate Nasal Spray
Started | 304 | 101
Completed | 285 | 92
Not Completed | 19 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dymista Nasal Spray | Fluticasone Propionate Nasal Spray | Total
Number analyzed (Participants) | 304 | 101 | 405
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 304 | 101 | 405
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (2.07) | 8.1 (1.94) | 8.1 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 49 | 170
  Male | 183 | 52 | 235
Region of Enrollment [Number; unit: participants]
  United States | 304 | 101 | 405

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Report
Description: reports of treatment emergent adverse events
Time Frame: 3 months of treatment
Measure: Number; unit: event
Arm/Group | Dymista Nasal Spray | Fluticasone Nasal Spray
Number analyzed (Participants) | 302 | 98
event | 124 | 37

ADVERSE EVENTS:
Arm/Group | Dymista Nasal Spray | Fluticasone Propionate Nasal Spray
Serious Adverse Events (participants affected / at risk) | 1/304 | 0/101
Other Adverse Events (participants affected / at risk) | 114/304 | 25/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dymista Nasal Spray (N=304) | Fluticasone Propionate Nasal Spray (N=101)
gastroenteritis elevated LFT (Gastrointestinal disorders) | 1 (1) | 0 (0) — one case of gastroenteritis ,patient with history of Chron's disease,deemed highly unlikely related to treatment, fully recovered
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dymista Nasal Spray (N=304) | Fluticasone Propionate Nasal Spray (N=101)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 | 9
headache (General disorders) | 20 | 3
cough (Respiratory, thoracic and mediastinal disorders) | 11 | 3
pyrexia (General disorders) | 10 | 2
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 0
otitis media (Ear and labyrinth disorders) | 9 | 3
vomiting (Gastrointestinal disorders) | 9 | 2
abdominal pain upper (Gastrointestinal disorders) | 8 | 2
upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Meda Pharmaceuticals requests that it receive copies of any intended communication at least 15 working days for an abstract or oral presentation and 45 working days for a manuscript). This is to allow Meda Pharmaceuticals to review the communications for accuracy , to verify that confidential information is not being inadvertently divulged, to provide any relevant supplementary information, and to allow establishment of co-authorship.